CLINICAL TRIAL: NCT02746978
Title: A Patient-centered Approach to Successful Community Transition After Catastrophic Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shepherd Center, Atlanta GA (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Michael Jones, Vice President Research and Technology, Shepherd Center, Atlanta GA
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IH-12-11-5106
Record Dates: First submitted 2016-02-29; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Spinal Cord Injury; Peer Group
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer directed education (Active Comparator): A revised education approach that focuses on problem solving discussions delivered by peers and grounded clinical information is compared to traditional approach of didactic clinician-driven education lectures
  Interventions: Other: Peer directed education
- Patient Engagement Portal (Other): A patient-owned portal to manage injury information is maintained in real-time by patients and families and shared with other care providers after inpatient rehabilitation discharge.
  Interventions: Other: Patient Engagement Portal

INTERVENTIONS:
Other: Peer directed education — No drug or device is included. The intervention of interest is the redesigned approach to inpatient education that follows the Stanford chronic disease self management approach which includes peer-led problem solving discussions compared to traditional didactic education lectures provided by nurse educators
  Arms: Peer directed education
Other: Patient Engagement Portal — No drug or device interventions. The Engagement Portal is populated by electronic medication record information (demographics, medications, supplies) then owned/maintained by patient after discharge. This approach to managing information and conditions associated with injury will be compared to the traditional approach of providing patients with a large instruction manual to carry home with them.
  Arms: Patient Engagement Portal

SUMMARY:
Shepherd Center is bringing a more patient-centered focus to educational, peer-support, and technology resources offered to patients with spinal cord injury and their families and is evaluating these changes.

Approximately 740 patients have provided information about healthcare utilization following inpatient rehabilitation. This information will help Shepherd Center staff follow utilization trends and plan programs targeted at the high-use areas.

DETAILED DESCRIPTION:
Research efforts are transforming the educational, peer-support and technology resources offered to patients and their caregivers, and evaluating how these changes help improve outcomes, including building patients' sense of self-efficacy - the belief that they can effectively manage their own care. Goals of the three focus areas include:

A. Patient and Family Education Revamp patient education modules for bladder management, skin management, and medical complications management to follow the chronic disease self management approach that replaces didactic lectures with participant-focused problem solving discussions led by peers (persons with SCI). Multiple baseline implementation approaches will be evaluated in interrupted time series analyses.

B. Peer mentoring and peer-led self-management training The peer mentor randomized clinical trial is reported separately on clinicaltrials.gov and not repeated here.

C. Patient and family web portal Shepherd Center, along with our collaborators at Craig Hospital in Denver, Colorado, are developing an engagement portal to provide a mechanism for patients to manage all aspects of injury following rehabilitation discharge and share information with other providers and caregivers.The portal will become a standard part of rehabilitation care and discharge planning for all Shepherd Center patients - starting first with patients with spinal cord injuries and later expanding to others. Stakeholders will be actively involved in providing feedback about portal usability and content so that the product continues to meet their needs.

ELIGIBILITY:
Inclusion Criteria:

* patient receiving inpatient rehabilitation at Shepherd Center following spinal cord injury
* discharge to community setting

Exclusion Criteria:

* discharge to non-community setting
* patient without spinal cord injury at Shepherd Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Rehospitalization | 30 days post rehabilitation discharge
  patient report on telephone interview

SECONDARY OUTCOMES:
Rehospitalization | 90 days post rehabilitation discharge
  patient report on telephone interview

OTHER OUTCOMES:
Depression as measured by the Patient Health Questionnaire (PHQ) | 180 days post rehabilitation discharge
  Data aggregated per scoring rules of validated measure. patient report on telephone interview
Societal participation as measured by CHART (Craig Handicap Assessment and Reporting Technique)- questionnaire | 180 days post rehabilitation discharge
  Data aggregated per scoring rules of validated measure. patient report on telephone interview
Satisfaction with Life Scale | 180 days post rehabilitation discharge
  patient report on telephone interview
Healthcare utilization - rehospitalization, emergency room visits, urgent care visits | 180 day post rehabilitation discharge
  per patient report on telephone interview
Press Gainey patient satisfaction with care - interview | 30 days post rehabilitation discharge
  Data aggregated per scoring rules of validated measure

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gassaway, Study Director — Dir Health and Wellness

IPD SHARING:
Plan to Share IPD: No